CLINICAL TRIAL: NCT03433833
Title: Phase 1 Study of Digoxin for Congenital Erythrocytosis Due to Up-Regulated Hypoxia Sensing
Brief Title: Digoxin for Congenital Erythrocytosis Due to Up-Regulated Hypoxia Sensing
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study Not Funded
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Victor Gordeuk, Professor of Medicine, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0064
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Polycythemia; Familial; Erythrocytosis; Familial; VHL Gene Mutation; HIF-2alpha Erythrocytosis; PHD2 Erythrocytosis; Chuvash Erythrocytosis
MeSH Terms: conditions — Polycythemia, primary familial and congenital | interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Patients will be given digoxin orally daily for 24 weeks. The initial dose will be selected with the goal of achieving a serum digoxin concentration of 0.5-0.9 ng/ml, a dose range recommended for heart failure patients. A dose of 0.0625, 0.125 or 0.25 mg daily will be selected based on a normogram.
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin — Digoxin oral route once daily for 24 weeks.
  Other Names: No other interventions

SUMMARY:
The investigators will study digoxin to inhibit the hypoxic response in congenital erythrocytosis due to germ line mutations that result in up-regulated hypoxia sensing. These forms of congenital erythrocytosis, characterized by augmented levels of hypoxia inducible factor (HIF)-1 and HIF-2, are due to mutations of VHL (von Hippel Lindau), EGLN1 (encoding prolyl hydroxylase 2 [PHD2]) and EPAS1 (endothelial PAS domain-containing protein 1) (encoding HIF-2α). In addition to a high hematocrit, patients have thrombotic complications and early mortality that are not improved by phlebotomy therapy. There is no effective therapy. Digoxin, long used to treat congestive heart failure, is a potent inhibitor of the master hypoxia-inducible transcription factor, HIF-1. The study hypothesis is that pharmacologic doses and levels of digoxin will decrease hemoglobin and hematocrit, decrease need for phlebotomy, decrease the propensity to thrombosis and decrease pulmonary pressure in patients with erythrocytosis due to up-regulated hypoxic responses. The clinical trial consists of 24 weeks of digoxin therapy in patients with hypoxic response-related erythrocytosis. The complete blood count, safety, symptoms of headache and lack of energy, echocardiogram, physical performance, and plasma products and blood cell expression of HIF-1-regulated genes are the outcome variables.

DETAILED DESCRIPTION:
The study will investigate digoxin to inhibit the hypoxic response in congenital erythrocytosis due to germ line mutations that result in up-regulated hypoxia sensing. These forms of congenital erythrocytosis, characterized by augmented levels of hypoxia inducible factor (HIF)-1 and/or HIF-2, are due to mutations of VHL (von Hippel Lindau), EGLN1 (encoding prolyl hydroxylase 2 [PHD2]) and EPAS1 (endothelial PAS domain-containing protein 1) (encoding HIF-2α). In addition to a high hematocrit, patients have thrombotic complications and early mortality that are not improved by phlebotomy therapy. There is no effective therapy. Digoxin, long used to treat congestive heart failure, is a potent inhibitor of the master hypoxia-inducible transcription factor, HIF-1, and likely HIF-2.

VHL mutations- 15 known patients in the US, 55 in Western Europe, 150 in Chuvashia, in Ischia and 11 in India.4 Chuvash erythrocytosis (CE), endemic in the Chuvash Republic of Russia and the Italian island of Ischia, is due to homozygosity for a missense mutation of VHL (VHL c.598C>T; VHL R200W). VHL R200W impairs interactions of VHL with HIF-α subunits, reducing their ubiquitin-mediated destruction. HIF-1 and HIF-2 heterodimers increase, leading to increased expression of their target genes, including erythropoietin (EPO). In addition, CE erythroid progenitors are hypersensitive to EPO, the explanation of which is not known. In pilot studies this hypersensitivity is inhibited by digoxin. CE patients are prone to develop thrombosis and early mortality that is independent of the increase in hematocrit. This phenotype is different from the dominantly inherited VHL tumor predisposition syndrome mutations that in combination with acquired somatic mutations result in tumorigenesis. Other homozygous and compound heterozygous VHL mutations that cause erythrocytosis but not tumors have been described.

EGLN1 (Egl-9 family hypoxia inducible factor 1) mutations- 5 patients in the US. and 21 in Europe. PHD2 (encoded by the EGLN1 gene) is, along with VHL, a principal negative regulator of HIFs. It targets HIF-α subunits for degradation. The first loss-of-function mutation of PHD2 (PHD2 P317R) was identified in a family in which heterozygotes had mild or borderline erythrocytosis. Since then, 25 additional patients with unexplained erythrocytosis who are heterozygote carriers of different PHD2 mutations have been reported. Almost all patients with PHD2-associated erythrocytosis have normal EPO levels.

EPAS1 mutations- 20 known patients in the US and approximately 100 in Europe. Affected patients have heterozygous missense mutations in the coding sequence of the EPAS1 gene encoding HIF-2α that result in gain-of function of HIF-2 and elevated EPO levels. There is heterogeneity in these gain-of-function EPAS1 mutations, but their existence supports the critical role of HIF-2 in controlling the expression of renal EPO.

Digoxin as an agent to inhibit HIFs. Digoxin, a common and readily available FDA-approved drug for treatment of congestive heart failure, was found to inhibit HIF-dependent gene transcription by ~90% at a concentration of 0.4 μM; it also inhibits HIF-1α protein translation and blocks HIF-1 activity in vivo. Doses of digoxin that prevent and treat murine hypoxic pulmonary hypertension partially protect from hypoxia-induced erythrocytosis. These doses lead to plasma digoxin levels in mice that are at or below the therapeutic range for humans. In unpublished data, therapeutic doses of digoxin diminished exaggerated erythropoiesis in vitro in a CE subject.

The study hypothesizes that pharmacologic doses and levels of digoxin will decrease hemoglobin and hematocrit, decrease need for phlebotomy, decrease the propensity to thrombosis and decrease pulmonary pressure in patients with erythrocytosis due to upregulated hypoxic responses. The proposed study is conducted under IND138480 and is approved by the FDA.

Aim 1. Determine if digoxin is safe and will decrease EPO, hemoglobin concentration and pulmonary pressure in patients with congenital erythrocytosis due to up-regulated hypoxia sensing.

Aim 2. Determine if digoxin will decrease purified blood cell lineage transcription and reduce plasma levels of the products of pro-thrombotic genes up-regulated by the hypoxic response, including IL1B (interleukin-1 beta), THBS1 (thrombospondin), EGR1 (early growth response 1), NLRP3 (NLR family pyrin domain containing 3), SERPINE1 (serpin family E member 1), and F3 (tissue factor).

Aim 3. In a corollary study, determine if in vivo achievable digoxin concentrations abrogate in vitro erythroid progenitor EPO hypersensitivity of mutations other than VHL R200W, and if HIF-2α inhibitors (already in clinical trials) abrogate erythroid progenitor EPO hypersensitivity alone or in combination with digoxin.

In summary, this proposal provides an unprecedented opportunity to identify inexpensive therapy for rare forms of erythrocytosis due to up-regulated hypoxia sensing for which there is now no safe, effective therapy. As such, this proposal fully coincides with the goals of the FDA's Orphan Products Program. The research will also help define the role of hypoxia in common maladies of mankind including chronic mountain sickness, obstructive sleep apnea, deep vein thrombosis, cancer associated thrombosis and pulmonary hypertension.

ELIGIBILITY:
Inclusion criteria. To be eligible to participate, an individual must meet all of the following criteria:

* Have mutation of VHL (von Hippel Lindau), EGLN1 (encoding prolyl hydroxylase 2 [PHD2]) or EPAS1 (encoding HIF-2α) that has been associated with congenital erythrocytosis with upregulated hypoxia sensing.
* Have an up-regulated hypoxic response defined by a hemoglobin concentration of greater than 15.5 g/dL in women and 17.5 g/dL in men in association with a serum EPO concentration that is increased above the reference range or that is in the reference range but above the expected level given the presence of erythrocytosis, i.e. above the lower quartile of the range.
* Male or female, aged 18 years and older.
* For females of reproductive potential: use of highly effective contraception for 1 month prior to screening and agreement to use such a method during study participation and for an additional two weeks after the end of digoxin administration.

Exclusion criteria. An individual who meets any of the following criteria will be excluded from participation:

* Diagnosis of polycythemia vera or high oxygen affinity hemoglobinopathy.
* End stage renal disease: estimated GFR <15 mL/min/1.73 m2 or receiving hemodialysis or peritoneal dialysis.
* Electrolyte imbalance: potassium <3.5 mEq/L, magnesium <1.8 mg/dL, or calcium >10.7 mg/dL.
* Hyperthyroidism (TSH <0.3 U/ml and T4 >12 μg/dL) or hypothyroidism (TSH > 6 U/ml).
* Myocarditis.
* History of hypersensitivity, arrhythmia or severe gastrointestinal side effects related to digoxin.
* Presence or history of any of the following conditions: first or second-degree AV block, Wolff-Parkinson-White Syndrome, other cardiac conduction abnormalities, or heart failure with preserved left ventricular systolic function including restrictive cardiomyopathy, constrictive pericarditis, amyloid heart disease, acute cor pulmonale and idiopathic hypertrophic subaortic stenosis.
* Peripheral arterial disease or ischemic heart disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin concentration | 24 weeks
  Change of 1.5 g/dL or more

SECONDARY OUTCOMES:
Serum EPO concentration | 24 weeks
  Change in log Epo concentration of 15% or more
Plasma concentration of PAI-1 (plasminogen activator inhibitor 1) | 24 weeks
  Change compared to baseline
Granulocyte mRNA (messenger ribonucleic acid) expression of F3 as determined by RT-PCR (reverse transcription polymerase chain reaction) | 24 weeks
  Change compared to baseline
Tricuspid regurgitation velocity determine by echocardiogram | 24 weeks
  Change compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Victor R Gordeuk, MD, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No
The research data will be shared with the co-investigators and the referring physicians.